CLINICAL TRIAL: NCT02729831
Title: Comparative Effectiveness of Decision Support Strategies for Joint Replacement Surgery: A Factorial Randomized Trial
Brief Title: Comparative Effectiveness of Decision Support Strategies for Joint Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Newton-Wellesley Hospital (Other); The New England Baptist Hospital (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director, Health Decision Sciences Center, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000229
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: decision making; decision aids; decision quality instruments; osteoarthritis; shared decision making
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Interactive Decision Aid and Usual Care (Experimental): Group receiving brief interactive decision aid and being seen by a provider assigned to usual care. The decision aids are the Shared Decision Points for hip and knee osteoarthritis from Healthwise.
  Interventions: Behavioral: Interactive decision aid
- Video decision aid and usual care (Experimental): Group receiving long video decision aids and being seen by a provider assigned to usual care. The decision aids are the DVD and Booklets for hip and knee osteoarthritis from Health Dialog.
  Interventions: Behavioral: Video decision aid
- Interactive Decision Aid and Provider Report (Experimental): Group receiving brief interactive decision aid and being seen by a provider assigned to intervention arm. The decision aids are the Shared Decision Points for hip and knee osteoarthritis from Healthwise. The provider intervention is a report that includes the patients' goals and treatment preferences.
  Interventions: Behavioral: Interactive decision aid; Behavioral: Provider Report
- Video decision aid and Provider report (Experimental): Group receiving long video decision aids and being seen by a provider assigned to intervention arm. The decision aids are the hip or knee DVD and Booklets for hip and knee osteoarthritis from Health Dialog. The intervention is a report that includes the patients' goals and treatment preferences.
  Interventions: Behavioral: Interactive decision aid; Behavioral: Provider Report

INTERVENTIONS:
Behavioral: Interactive decision aid — The Healthwise Shared Decision Points in booklet version for hip and knee osteoarthritis
  Arms: Interactive Decision Aid and Provider Report; Interactive Decision Aid and Usual Care; Video decision aid and Provider report
Behavioral: Video decision aid — Health Dialog DVD and booklet decision aids for hip and knee osteoarthritis
  Arms: Video decision aid and usual care
Behavioral: Provider Report — A short report that includes the patients' goals and treatment preferences
  Arms: Interactive Decision Aid and Provider Report; Video decision aid and Provider report

SUMMARY:
This study is a 2X2 factorial randomized trial that will the examine the comparative effectiveness of two patient decision aids for hip and knee osteoarthritis (OA) as well as the impact of a surgeon-focused intervention.

DETAILED DESCRIPTION:
This study is a 2X2 factorial randomized trial that will examine the comparative effectiveness of different decision support strategies for patients making treatment decisions about hip or knee osteoarthritis (OA). Eligible patient subjects will be randomly assigned to receive one of two decision aids before their upcoming clinic visit with a participating orthopedic specialist. Participating providers are randomly assigned to either usual care or an intervention (a report that includes patients' goals and treatment preferences). Patient participants will complete three surveys at different time points: before their orthopedic visit, one week after the clinic visit, and 12 months later. Providers will complete a short survey for a subset of patient participants. The study is titled the DECIDE-OA study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either hip or knee osteoarthritis
* Scheduled visit with participating orthopedic surgeon

Exclusion Criteria:

* prior partial or total knee or hip joint replacement within last 5 years
* hip fracture or asceptic necrosis (AVN) in last 12 months
* Rheumatoid arthritis
* Psoriatic arthritis
* Unable to read English or Spanish
* Unable to consent for self due to cognitive or medical issue
* Hip or knee decision aid provided by Partners Healthcare clinician within 12 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, de-identified copy of the final data set that includes survey data for the primary and secondary outcomes from patient participants has been created. The PI will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital (MGH) policies for data sharing. Investigators from other sites are able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team, etc.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available September 2019 and will be available for at least 7 years from that time.
Access Criteria: Interested investigators may consult the DECIDE-OA study page on the Massachusetts General Hospital's Health Decision Sciences Center website for information about data sharing.
URL: https://www.mghdecisionsciences.org

REFERENCES:
- [Background] Sepucha K, Feibelmann S, Chang Y, Clay CF, Kearing SA, Tomek I, Yang T, Katz JN. Factors associated with the quality of patients' surgical decisions for treatment of hip and knee osteoarthritis. J Am Coll Surg. 2013 Oct;217(4):694-701. doi: 10.1016/j.jamcollsurg.2013.06.002. Epub 2013 Jul 25. PMID 23891070
- [Background] Mangla M, Bedair H, Chang Y, Daggett S, Dwyer MK, Freiberg AA, Mwangi S, Talmo C, Vo H, Sepucha K. Protocol for a randomised trial evaluating the comparative effectiveness of strategies to promote shared decision making for hip and knee osteoarthritis (DECIDE-OA study). BMJ Open. 2019 Feb 24;9(2):e024906. doi: 10.1136/bmjopen-2018-024906. PMID 30804032
- Available data/document: outcome measure — https://mghdecisionsciences.org/tools-training/decision-quality-instruments/ — Hip Osteoarthritis Decision Quality Instrument
- Available data/document: outcome measure — https://mghdecisionsciences.org/tools-training/decision-quality-instruments/ — Knee Osteoarthritis Decision Quality Instrument

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2016-December 2017. Adults diagnosed with hip or knee osteoarthritis who had a visit scheduled with a participating orthopedic surgeon at 3 sites were invited to participate before their visit.
Pre-assignment Details: Participants were randomized to a study arm after screening the surgeons' schedules. To be eligible for the study, patients needed to attend the visit with the surgeon. The majority of post randomization exclusions are due to patients not showing up to the visit. Some are due to limited clinical information available at screening.
Period: Baseline (Post Decision Aid, Pre-visit)
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Started | 320 | 315 | 293 | 292
Completed | 282 | 292 | 275 | 275
Not Completed | 38 | 23 | 18 | 17
Not completed — Ineligible post completion | 38 | 23 | 18 | 17
Period: 1 Week Post-visit
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Started | 282 | 292 | 275 | 275
Completed | 239 | 252 | 237 | 239
Not Completed | 43 | 40 | 38 | 36
Not completed — Lost to Follow-up | 43 | 40 | 38 | 36
Period: 6 Month Follow-up
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Started (Follow-up survey (Period 3) was sent to all those who completed the Baseline (Period 1) survey.) | 282 | 292 | 275 | 275
Completed | 227 | 238 | 227 | 232
Not Completed | 55 | 54 | 48 | 43
Not completed — Lost to Follow-up | 54 | 51 | 48 | 42
Not completed — Death | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who attended a visit with an orthopedic surgeon, completed a Baseline survey, and subsequently remained clinically eligible post-visit. Study staff reviewed patient medical record post-visit to finalize enrollment in study, as limited data pre-visit meant there were some post-randomization exclusions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report | Total
Number analyzed (Participants) | 282 | 292 | 275 | 275 | 1124
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.6) | 64.6 (9.9) | 64.3 (10.3) | 64.9 (9.5) | 64.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 179 | 173 | 141 | 645
  Male | 130 | 113 | 102 | 134 | 479
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 13 | 5 | 3 | 24
  Not Hispanic or Latino | 230 | 235 | 227 | 229 | 921
  Unknown or Not Reported | 49 | 44 | 43 | 43 | 179
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 3 | 4 | 2 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  Black or African American | 6 | 8 | 1 | 4 | 19
  White | 258 | 261 | 255 | 243 | 1017
  More than one race | 3 | 5 | 4 | 4 | 16
  Unknown or Not Reported | 11 | 12 | 13 | 16 | 52
Joint [Count of Participants; unit: Participants] — Diagnosis of hip or knee osteoarthritis. Dx status collected from visit note and/or confirmed via x-ray report.
  Participants
    Hip | 85 | 79 | 95 | 108 | 367
    Knee | 197 | 213 | 180 | 167 | 757
Decision aid delivery [Count of Participants; unit: Participants] — Mode of delivery for the patient decision aid (DA). Participants who were registered users for the online Patient Gateway platform were sent the DA online to their account; all other patients were mailed a paper version.
  Participants
    Paper | 225 | 232 | 218 | 217 | 892
    Online | 57 | 60 | 57 | 58 | 232
Health literacy [Count of Participants; unit: Participants] — Single item literacy screener. One question assessing how often patients need help reading and understanding medical paperwork. Patient self-reported at T2 (pre-visit) survey.
  Participants
    Never | 191 | 197 | 197 | 197 | 782
    Rarely | 43 | 52 | 42 | 44 | 181
    Sometimes | 30 | 24 | 24 | 18 | 96
    Often | 6 | 10 | 3 | 7 | 26
    Always | 8 | 5 | 5 | 7 | 25
    Missing | 4 | 4 | 4 | 2 | 14
Education [Count of Participants; unit: Participants] — One question assessing highest level of education achieved. Patient self-reported at T2 (post-visit) survey.
  Participants
    8th grade or less | 4 | 3 | 1 | 2 | 10
    Some high school but did not graduate | 1 | 3 | 2 | 3 | 9
    High school graduate or GED | 31 | 38 | 26 | 22 | 117
    Some college or 2-year degree | 54 | 60 | 47 | 47 | 208
    4-year college graduate | 45 | 55 | 59 | 53 | 212
    More than a 4-year college degree | 101 | 89 | 98 | 105 | 393
    Missing | 46 | 44 | 42 | 43 | 175
Insurance [Count of Participants; unit: Participants] — Primary insurance type. Information collected from patient medical record.
  Participants
    Medicare | 81 | 93 | 68 | 79 | 321
    Medicaid/Dual eligible | 41 | 30 | 19 | 25 | 115
    Commercial | 109 | 119 | 93 | 80 | 401
    Missing | 51 | 50 | 95 | 91 | 287
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) calculated as a function of weight (kg)/height squared (m2). Information collected from patient medical record.
  kg/m^2 | 31.4 (6.8) | 30.9 (6.3) | 28.9 (6.4) | 29.7 (6.3) | 30.1 (6.5)
Charlson co-morbidity index (CCI) [Count of Participants; unit: Participants] — A summary score representing the burden of disease for a patient. A total of 18 comorbidities, with subcategories for diabetes, liver disease, and cancer were collected from the medical record. Each comorbidity is assigned a score from 1 to 6 based on mortality risk and disease severity, then summed to form the total CCI score (0 minimum score - 39 maximum score). Higher scores indicate higher mortality and burden of disease.
  Participants
    0 | 205 | 217 | 201 | 203 | 826
    1 | 33 | 38 | 36 | 35 | 142
    2 | 33 | 21 | 24 | 28 | 106
    3+ | 10 | 14 | 12 | 8 | 44
    Missing | 1 | 2 | 2 | 1 | 6
Quality of life (EQ-5D) [Mean (Standard Deviation); unit: units on a scale] — 5 item summary measure of overall health status. It generates a single index value, that ranges from best health 1 to worst health -0.11.
  units on a scale | 0.63 (0.19) | 0.62 (0.21) | 0.65 (0.20) | 0.65 (0.18) | 0.64 (0.20)

OUTCOME MEASURES:

1. Primary Outcome: Patients Knowledge
Description: Knowledge sub-score generated from responses to the Hip or Knee Decision Quality Instrument (DQI). Scores range from 0-100%, with higher score meaning higher knowledge.
Time Frame: before orthopedic visit
Population: There were a total of 5 hip and knee specific knowledge questions in the DQI. Participants must answer at least 3 out of 5 questions to get a total knowledge score out of 100%. Only 1082/1124 participants provided sufficient information to calculate a knowledge score.
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Number analyzed (Participants) | 274 | 276 | 268 | 264
percentage of correct answers | 79 (25) | 71 (24) | 84 (21) | 75 (23)
Statistical Analysis 1: Comparison: Interactive Decision Aid and Usual Care vs Video Decision Aid and Usual Care vs Interactive Decision Aid and Provider Report vs Video Decision Aid and Provider Report; The comparison groups were: Interactive decision versus Video decision aid; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = 9, 95% CI 2-sided [6 to 12]

2. Primary Outcome: Percentage of Patients Who Received Preferred Treatment
Description: Patient preferred treatment item from the Hip or Knee Decision Quality Instrument will be compared with the treatment received to determine percentage of patients who received treatment that matched their preferences.
Time Frame: 1 week after visit with orthopedic surgeon
Population: Participants must complete the 1 week survey and answer the treatment preference question. Only 956/967 participants provided sufficient information to calculate a treatment match.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Number analyzed (Participants) | 237 | 249 | 232 | 238
Participants | 175 | 182 | 166 | 177
Statistical Analysis 1: Comparison: Interactive Decision Aid and Usual Care vs Video Decision Aid and Usual Care vs Interactive Decision Aid and Provider Report vs Video Decision Aid and Provider Report; We tested for interaction effects. Comparison groups were: MD Usual Care vs. MD Provider report; Test type: Superiority; p = 0.86, Regression, Logistic; General Estimating Equations accounted for clustering of patients within surgeons and controlling for baseline EQ-5D, BMI, joint and education; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.74 to 1.44]
Statistical Analysis 2: Comparison: Interactive Decision Aid and Usual Care vs Video Decision Aid and Usual Care vs Interactive Decision Aid and Provider Report vs Video Decision Aid and Provider Report; We tested for interaction effects. Comparison groups are: Interactive decision versus Video decision aid; Test type: Superiority; p = 0.75, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.76 to 1.47]

3. Secondary Outcome: Percentage of Participants Who Used the Decision Aid
Description: 1 item asking patients how much they reviewed the program (none, some, most, all). The percentage who report viewing most or all will be calculated.
Time Frame: before orthopedic visit
Population: Participants must answer the program usage question on the Baseline survey. Only 1091/1124 participants provided sufficient information to calculate decision aid usage.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Number analyzed (Participants) | 277 | 283 | 262 | 269
Participants
  None | 42 | 38 | 27 | 34
  Some | 38 | 45 | 32 | 42
  Most | 24 | 68 | 24 | 66
  All | 173 | 132 | 179 | 127
Statistical Analysis 1: Comparison: Interactive Decision Aid and Usual Care vs Video Decision Aid and Usual Care vs Interactive Decision Aid and Provider Report vs Video Decision Aid and Provider Report; Comparison groups were: patients who reported using all of the DA versus everyone else; Test type: Superiority; p < 0.001, Chi-squared; Compared patients who reported using all of the DA compared to everyone else; Risk Difference (RD) = 18.5, 95% CI 2-sided [12.8 to 24.5]

4. Secondary Outcome: Change in Quality of Life
Description: Overall quality of life (EQ-5D) scores will be calculated and the impact of decision support strategies on change in quality of life will be examined. Scale ranges from -0.11 to 1.00, with higher (positive) values meaning better overall health. The minimum important change is 0.10 points.
Time Frame: before orthopedic visit; 12 months from date of orthopedic visit
Population: Participants must answer all 5 items of the EQ-5D measure from the Baseline and 6 months follow-up survey. Only 868/1124 participants provided sufficient information at both time points to calculate a change in quality of life score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Number analyzed (Participants) | 212 | 224 | 215 | 217
units on a scale | 0.17 (0.21) | 0.15 (0.22) | 0.15 (0.23) | 0.16 (0.20)
Statistical Analysis 1: Comparison: Interactive Decision Aid and Usual Care vs Video Decision Aid and Usual Care vs Interactive Decision Aid and Provider Report vs Video Decision Aid and Provider Report; We included all 4 study groups, but the comparison group was: informed, patient centered decision yes vs. no; Test type: Superiority; p < 0.001, Regression, Linear; Generalized Estimating Equation accounting for clustering within surgeons. Model included treatment, sex, age, education, site and joint; Mean Difference (Net) = 0.04, 95% CI 2-sided [0.016 to 0.065]

5. Secondary Outcome: Surgical Rates
Description: Medical chart review and patient report of whether or not surgery was used in the 6 months after the visit.
Time Frame: 6 months after the initial visit
Population: Excluding patients who did not provide information to calculate the Informed, Patient-Centered (IPC) variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
Number analyzed (Participants) | 239 | 252 | 237 | 239
Participants | 140 | 153 | 134 | 154
Statistical Analysis 1: Comparison: Interactive Decision Aid and Usual Care vs Video Decision Aid and Usual Care vs Interactive Decision Aid and Provider Report vs Video Decision Aid and Provider Report; We included all 4 study groups, but the comparison group was: informed, patient centered (IPC) decision yes vs. no. We excluded those who did not provide information to calculate the IPC variable; Test type: Superiority; p < 0.001, Regression, Logistic; General estimating equations were used to account for clustering of patients within surgeons; Odds Ratio (OR) = 25.7, 95% CI 2-sided [16.5 to 40.1]

ADVERSE EVENTS:
Time Frame: The 1 week post visit and 6 month follow-up surveys were checked as they came in for evidence of adverse events.
Arm/Group | Interactive Decision Aid and Usual Care | Video Decision Aid and Usual Care | Interactive Decision Aid and Provider Report | Video Decision Aid and Provider Report
All-Cause Mortality (participants affected / at risk) | 0/282 | 0/292 | 0/275 | 0/275
Serious Adverse Events (participants affected / at risk) | 0/282 | 0/292 | 0/275 | 0/275
Other Adverse Events (participants affected / at risk) | 0/282 | 0/292 | 0/275 | 0/275

LIMITATIONS AND CAVEATS:
Study staff and participating surgeons not blinded to intervention; 6 months may be too short to capture full benefit of surgery on quality of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02729831/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02729831/SAP_001.pdf